CLINICAL TRIAL: NCT06096961
Title: The Effect Of Baby Smell On The Amount Of Breast Milk, Salivary Cortisol Level And Mother Baby Attachment: A Randomized Controlled Study
Brief Title: The Effect Of Baby Smell On The Amount Of Breast Milk, Salivary Cortisol Level And Mother Baby Attachment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Öykü Bali, Principal Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: OYKUCALISMA
Record Dates: First submitted 2023-10-04; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Mother-Infant Interaction; Premature Birth
Keywords: mother milk; stress; mother baby bonding; premature
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: There are two groups in the study: experimental and control groups. Mothers in the experimental group will be given baby clothes that their babies will wear for 12 hours and will be asked to smell these clothes during the milking process. The work will continue for four days. Mothers in the intervention group will smell their baby's scented diapers, and mothers in the control group will express their milk without any intervention and record the amount.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mothers using baby scent (Experimental): Mothers in the experimental group will be given baby clothes that their babies will wear for 12 hours and will be asked to smell these clothes during the milking process. The work will continue for four days. Saliva cortisol test and mother-infant attachment scale will be applied on the first day and the last day.
  Interventions: Behavioral: Baby smell
- Mothers who do not use baby scent (No Intervention): Mothers in the control group will express milk without any intervention. The works will continue for 4 days. Saliva cortisol test and mother-baby attachment scale will be applied on the first day and the last day.

INTERVENTIONS:
Behavioral: Baby smell — Mothers in the experimental group will be given baby clothes that their babies will wear for 12 hours and will be asked to smell these clothes during the milking process.
  Arms: Mothers using baby scent

SUMMARY:
The goal of this [type of study: randomized controlled clinical trial] is to [determine the effect of applying the scent of premature newborns who cannot be breastfed to the mother on the mother's milk amount, salivary cortisol level and mother-infant attachment.] in [mothers of premature babies]. The main question[s] it aims to answer are:

* [Hypothesis 1: There is a difference in the amount of milk of the mother.]
* [Hypothesis 2: There is a difference in the level of cortisol in the mother's saliva.]
* [Hypothesis 3: There is a difference in terms of mother-baby attachment level.] Participants will [Participants will express milk and record the amount of milk.].

If there is a comparison group: Researchers will compare [control and experimental groups] to see if [difference in amount of milk, cortisol level, baby attachment].

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study to determine the effect of applying the scent of non-breastfeedable premature newborns to the mother on the mother's milk quantity, salivary cortisol level and mother-baby bonding. The study is planned to be conducted with the mothers of premature infants whose babies are hospitalized in the Neonatal Intensive Care Unit of Bursa City Hospital. There will be two groups in the study: study and control group. For each group, 30 mothers will be included in the study. The study will continue for four days. The mothers in the experimental group will be given the gowns that their babies wear for 12 hours and they will be asked to smell these gowns during the milking process. On the 1st day, mothers in both groups will be trained on expressing and storing breast milk (frequency of expressing milk, appropriate speed of the pump, milk storage bags, room temperature, storage times in the refrigerator and freezer). All mothers will be ensured to express their milk with the same milk pumps. Mothers will be provided with a syringe to measure their milk. The mothers will be asked to express their milk at three-hour intervals and record the amount measured. Mothers in the experimental group will be asked to smell their babies' scented clothes during the milking process. A sample will be taken from the mothers to look at the cortisol level in saliva. Data collection forms will be filled in. On the 2nd and 3rd day, mothers will be asked to express their milk at three-hour intervals and record the amount they measured on the mother follow-up form. The mothers in the experimental group will be asked to smell their babies' smelly clothes during the milking process. On the 4th day, mothers will be asked to express their milk at three-hour intervals and record the amount they measured on the mother follow-up form. The mothers in the experimental group will be asked to smell their babies' scented clothes during the milking process. The mothers will be sampled again to check the cortisol level in saliva. Mother-infant attachment scale will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Mother's acceptance of the application
* Ability to communicate with the mother (being literate, speaking Turkish, etc.)
* Gestational week being 34 weeks or less
* The newborn is in the NICU

Exclusion Criteria:

* The newborn's gestational age is over 34 weeks
* The mother is breastfeeding her baby
* Being a smoker (Ahmed et al. 2019)
* The mother is unable to express milk due to a serious chronic disease or pregnancy complication.
* The mother has a breast problem that may affect milk expression (cracked, mastitis, collapse, etc.).
* If the mother uses milk-boosting drinks or food

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only mothers can participate in the study.
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
amount of breast milk | Mothers participating in the study will express their milk every three hours for four days and record the amount of milk.

SECONDARY OUTCOMES:
mother baby attachment scale | The mother-infant attachment scale will be applied to the mothers participating in the study on the first and fourth day of the study.
  This scale, which can be applied from the first day after birth and shows the relationship between the mother's mood and the bond established, allows the mother to express the feelings she feels towards her baby with a single word. The scale, whose original name is "Mother-to-Infant Bonding Scale", was developed by Taylor et al. in 2005. It was adapted into Turkish by Aydemir and Alparslan (2008). The scale is a 4-point Likert type and consists of eight items. Responses consist of four options and are scored between 0 and 3. Since they express positive emotion, the first, fourth and sixth items are scored as 0, 1, 2, 3, and since they express negative emotion, the second, third, fifth, seventh and eighth items are scored as 3, 2, 1, 0. The lowest score that can be obtained is 0, the highest score is 24.
salivary cortisol level | Saliva cortisol test will be applied to the mothers participating in the study on the first and fourth day of the study.

CONTACTS AND LOCATIONS:
Overall Officials: AYFER ACIKGOZ, Study Director — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akkoca Z, Yigit D, Acikgoz A. The Effect of Neonates' Exposure to Their Mother's Scent on Weight Gain: A Randomized Controlled Study. Breastfeed Med. 2022 Jan;17(1):79-84. doi: 10.1089/bfm.2021.0274. Epub 2021 Dec 22. PMID 34939823
- [Background] Cakirli M, Acikgoz A. A Randomized Controlled Trial: The Effect of Own Mother's Breast Milk Odor and Another Mother's Breast Milk Odor on Pain Level of Newborn Infants. Breastfeed Med. 2021 Jan;16(1):75-81. doi: 10.1089/bfm.2020.0222. Epub 2020 Oct 20. PMID 33085532
- [Background] Chrustek A, Dombrowska-Pali A, Olszewska-Slonina D. Analysis of the composition and antioxidant status of breast milk in women giving birth prematurely and on time. PLoS One. 2021 Jul 23;16(7):e0255252. doi: 10.1371/journal.pone.0255252. eCollection 2021. PMID 34297788
- [Background] Holditch-Davis D, Santos H, Levy J, White-Traut R, O'Shea TM, Geraldo V, David R. Patterns of psychological distress in mothers of preterm infants. Infant Behav Dev. 2015 Nov;41:154-63. doi: 10.1016/j.infbeh.2015.10.004. Epub 2015 Oct 22. PMID 26495909
- [Background] Ak J, Lakshmanagowda PB, G C M P, Goturu J. Impact of music therapy on breast milk secretion in mothers of premature newborns. J Clin Diagn Res. 2015 Apr;9(4):CC04-6. doi: 10.7860/JCDR/2015/11642.5776. Epub 2015 Apr 1. PMID 26023551
- [Background] Miller J, Tonkin E, Damarell RA, McPhee AJ, Suganuma M, Suganuma H, Middleton PF, Makrides M, Collins CT. A Systematic Review and Meta-Analysis of Human Milk Feeding and Morbidity in Very Low Birth Weight Infants. Nutrients. 2018 May 31;10(6):707. doi: 10.3390/nu10060707. PMID 29857555
- [Background] Montirosso R, Provenzi L, Calciolari G, Borgatti R; NEO-ACQUA Study Group. Measuring maternal stress and perceived support in 25 Italian NICUs. Acta Paediatr. 2012 Feb;101(2):136-42. doi: 10.1111/j.1651-2227.2011.02440.x. Epub 2011 Sep 14. PMID 21827551
- [Background] Neu M, Hazel NA, Robinson J, Schmiege SJ, Laudenslager M. Effect of holding on co-regulation in preterm infants: a randomized controlled trial. Early Hum Dev. 2014 Mar;90(3):141-7. doi: 10.1016/j.earlhumdev.2014.01.008. Epub 2014 Jan 27. PMID 24480604
- [Background] Rojas MA, Kaplan M, Quevedo M, Sherwonit E, Foster L, Ehrenkranz RA, Mayes L. Somatic growth of preterm infants during skin-to-skin care versus traditional holding: a randomized, controlled trial. J Dev Behav Pediatr. 2003 Jun;24(3):163-8. doi: 10.1097/00004703-200306000-00006. PMID 12806228
- [Background] Tasci B, Kuzlu Ayyildiz T. The Calming Effect of Maternal Breast Milk Odor on Term Infant: A Randomized Controlled Trial. Breastfeed Med. 2020 Nov;15(11):724-730. doi: 10.1089/bfm.2020.0116. Epub 2020 Oct 29. PMID 33121256
- [Background] Taylor A, Atkins R, Kumar R, Adams D, Glover V. A new Mother-to-Infant Bonding Scale: links with early maternal mood. Arch Womens Ment Health. 2005 May;8(1):45-51. doi: 10.1007/s00737-005-0074-z. Epub 2005 May 4. PMID 15868385
- [Background] Trend S, Strunk T, Lloyd ML, Kok CH, Metcalfe J, Geddes DT, Lai CT, Richmond P, Doherty DA, Simmer K, Currie A. Levels of innate immune factors in preterm and term mothers' breast milk during the 1st month postpartum. Br J Nutr. 2016 Apr 14;115(7):1178-93. doi: 10.1017/S0007114516000234. Epub 2016 Feb 19. PMID 26891901
- [Background] Ahmed, F., Jean-Baptiste, F., Thompson, A., Nwokorie, U., Nya, G. E., & Bassey, G. O. . Effects of maternal tobacco smoking on breast milk composition and infant development: a literature review. J Bacteriol Mycol Open Access. 2019; 7(5): 107-110.
- [Background] Aydemir Karakulak, H, Alparslan, Ö. Anne-bebek bağlanma ölçeğinin türk toplumuna uyarlanması: Aydın örneği . Çağdaş Tıp Dergisi. 2016; 6 (3) : 188-199 .
- [Background] Dabas S, Joshi P, Agarwal R, Yadav RK, & Kachhawa G. Impact of audio assisted relaxation technique on stress, anxiety and milk output among postpartum mothers of hospitalized neonates: A randomized controlled trial. Journal of Neonatal Nursing. 2019; 25(4): 200-204.
- [Background] De Clifford-Faugère G, Aita M, Héon M,& Le May S. Management of procedural pain in preterm infants through olfactive stimulation with mothers' milk: A pilot study. Science of Nursing and Health Practices. 2019; 2(1): 1-13.
- [Background] Kömürcü B. Erken doğan bebek annelerinde travma sonrası stres: ilişkili etmenler ve müdahale çalışmaları üzerine bir derleme. Nesne-Psikoloji Dergisi. 2020; 8(16): 158-170.
- [Background] Merter ÖS, Altay N. Yenidoğan yoğun bakımda izlenen prematüre bebeklerin anne sütü ile beslenme durumlarının değerlendirilmesi. Gazi Sağlık Bilimleri Dergisi. 2020; 5 (1): 21-29.
- [Background] Özlü F, Tunç A, Yıldızdaş HY, & Büyükkurt S. Geç prematüre doğan bebeklerin postnatal ilk 15 günde karşılaştıkları sorunların değerlendirilmesi. Çocuk Sağlığı ve Hastalıkları Dergisi. 2017; 60(2): 39-54.
- [Background] Suzan ÖK. Kolostrum: Özellikleri ve prematüre bebeğe faydaları. Sürekli Tıp Eğitimi Dergisi. 2020; 29(3): 221-227
- [Background] Varışoğlu Y, Güngör Satılmış İ. Preterm doğumlarda anne sütü ve anne sütünü artırmaya yönelik alternatif yöntemler . Izmir Democracy University Health Sciences Journal. 2019; 2 (2): 99-113 .
- See also: Related Info — https://www.who.int/publications/i/item/9789240005648
- See also: Related Info — https://www.who.int/news-room/fact-sheets/detail/preterm-birth
- See also: Related Info — https://www.resmigazete.gov.tr/eskiler/2011/04/20110419-5.htm
- Available data/document: thesis — http://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp — Kara, A. (2022). Bebekleri yenidoğan yoğun bakım ünitesi'nde yatan annelerde bebek kokusunun anksiyete ve süt miktarına etkisi [Yüksek Lisans Tezi, Marmara Üniversitesi Sağlık Bilimleri Enstitüsü]. YÖK Ulusal Tez Merkezi.
- Available data/document: thesis — http://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp — Turhan İ. (2020). Bebeği yenidoğan ünitesinde yatan annelere bebeğinin video görüntüsünün izletilmesinin anne sütü ve maternal bağlanmaya etkisi [Yüksek Lisans Tezi, Erciyes Üniversitesi Sağlık Bilimleri Enstitüsü]. YÖK Ulusal Tez Merkezi.
- Available data/document: thesis — http://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp — Varişoğlu, Y. (2019). Yenidoğan yoğun bakım ünitesinde prematüre bebeği olan annelere dinletilen müziğin anne sütü üretimine etkisi. [Doktora Tezi, İstanbul Üniversitesi Cerrahpaşa Lisansüstü Eğitim Enstitüsü]. YÖK Ulusal Tez Merkezi.